CLINICAL TRIAL: NCT01925235
Title: Remote Ischemic Preconditioning Effects on Kidney Function in Patients Receiving Transcatheter Aortic Valve Implantation
Brief Title: Analysis of Remote-ischemic Preconditioning Effects on Kidney Function
Acronym: RenPRO-TAVI
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Fikret Er, Associate Professor, University of Cologne
Other Study IDs: Ren-PRO TAVI retro
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Renal Function; Renal Injury
Keywords: remote ischemic preconditioning; acute kidney injury; TAVI; RenPRO trial; parameters
MeSH Terms: conditions — Acute Kidney Injury | interventions — Inflation, Economic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: patients with impaired renal function and a high risk of developing acute kidney injury undergoing TAVI and receiving standard care including pre-hydration 12 hours prior and 12 hours post procedure
- RIPC: patients with impaired renal function and a high risk of developing acute kidney injury undergoing TAVI and receiving standard care including pre-hydration 12 hours prior and 12 hours post procedure plus ischemic preconditioning (intermittent arm ischemia through 4 cycles of 5-minute inflation and 5-minute deflation of a blood pressure cuff)
  Interventions: Procedure: remote ischemic preconditioning

INTERVENTIONS:
Procedure: remote ischemic preconditioning
  Other Names: intermittent arm ischemia through 4 cycles of 5-minute inflation and 5-minute deflation of a blood pressure cuff
  Groups: RIPC

SUMMARY:
Patients with impaired renal function are at elevated risk for development of acute kidney injury (AKI). AKI is associated with increased risk for cardiovascular morbidity and mortality. Effective AKI prevention strategies are needed. Remote ischemic preconditioning (RIPC) is a novel and successful strategy to attenuate contrast medium induced AKI in patients undergoing elective coronary angiography.

The retrospective RenPro-TAVI Trial was designed to test the hypothesis whether remote ischemic preconditioning might attenuate kidney injury in patients receiving transcatheter aortic valve implantation (TAVI).

Patients with impaired renal function undergoing TAVI will be evaluated in respect whether they received remote ischemic preconditioning before the procedure or not. This study will give insight if RIPC might be beneficial in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* impaired renal function (baseline eGFR of <60 ml/min)
* high INTEGER risk score > 11
* high EuroSCORE (European system for cardiac operative risk evaluation)

Exclusion Criteria:

* severe renal impairment (eGFR <15 ml/min and/or in chronic dialysis)
* recent (<=30 days) contrast media exposure
* patients enrolled in concomitant studies
* fertile women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with impaired renal function and a high risk of developing contrast medium-induced acute kidney injury undergoing TAVI
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
change in parameters determining renal function and injury | 48 hours after TAVI
  serum creatinine, cystatin c, urinary neutrophil gelatinase-associated lipocalin (NGAL)

SECONDARY OUTCOMES:
acute kidney injury | 48 hours after TAVI
  increase in serum creatinine ≥25% or ≥0.5 mg/dL above baseline at 48 hours after TAVI

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Er F, Nia AM, Dopp H, Hellmich M, Dahlem KM, Caglayan E, Kubacki T, Benzing T, Erdmann E, Burst V, Gassanov N. Ischemic preconditioning for prevention of contrast medium-induced nephropathy: randomized pilot RenPro Trial (Renal Protection Trial). Circulation. 2012 Jul 17;126(3):296-303. doi: 10.1161/CIRCULATIONAHA.112.096370. Epub 2012 Jun 26. PMID 22735306
- [Background] Er F, Nia AM, Dopp H, Dahlem KM, Caglayan E, Erdmann E, Gassanov N, Hellmich M, Burst V, Kubacki T, Benzing T. Response to letter regarding article, "Ischemic preconditioning for prevention of contrast medium-induced nephropathy: randomized Pilot RenPro-Trial (Renal Protection Trial)". Circulation. 2013 Apr 2;127(13):e536. doi: 10.1161/circulationaha.112.147587. No abstract available. PMID 23662313
- See also: Related Info — http://www.cardiovascular-research.org